CLINICAL TRIAL: NCT01676649
Title: A Phase II Study of Ipilimumab in Combination With Carboplatin and Paclitaxel in Patients With Unresectable Stage III or Stage IV Melanoma
Brief Title: Ipilimumab With Carboplatin and Paclitaxel in Patients With Unresectable Stage III and Stage IV Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Wilson Miller, Medical Oncologist, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-195
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Untreated Stage III Melanoma or Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Arm A: Carboplatin (week 1, week 4, week 7, week 10, and week 13) Paclitaxel (week 1, week 4, week 7, week 10, and week 13) Ipilimumab (week 4, week 7, week 10, and week 13)
  Interventions: Biological: Ipilimumab; Drug: Carboplatin; Drug: Paclitaxel
- B (Experimental): Carboplatin (week 1, week 4, week 7, week 10, and week 13) Paclitaxel (week 1, week 4, week 7, week 10, and week 13) Ipilimumab (week 5, week 8, week 11, and week 14)
  Interventions: Biological: Ipilimumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: Ipilimumab — 3 mg/kg
  Other Names: YERVOY
Drug: Carboplatin — AUC = 6
Drug: Paclitaxel — 175 mg/m2

SUMMARY:
The safety of the combination of ipilimumab with carboplatin/paclitaxel treatment with two different dosing schedules will be investigated in patients with metastatic melanoma. This protocol will also investigate both the clinical benefit of this combination and the features of the host immune system that may predict response to ipilimumab with chemotherapy in patients with unresectable Stage III and Stage IV melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent.
* Histologic diagnosis of malignant melanoma
* Untreated unresectable Stage III melanoma with N3 macroscopic lymph nodes or in-transit/satellite metastases or Stage IV melanoma (note that prior adjuvant melanoma therapy is permitted). Prior treatment with BRAF inhibitors in the metastatic setting is also permitted.
* Measurable/evaluable disease
* Required values for initial laboratory tests:

  * WBC ≥ 2000/uL
  * ANC ≥ 1.5 x 10E9/L
  * Platelets ≥ 100 x 10E9/L
  * Hemoglobin ≥ 90 g/L (may be transfused)
  * Creatinine Clearance ≥ 50 ml/min (calculated -Cockcroft-Gault)
  * AST/ALT ≤ 2.5 x ULN for patients without liver metastasis,

    ≤ 5 times for liver metastases
  * Bilirubin ≤ 2.5 x ULN
* No active or chronic infection with HIV, Hepatitis B, or Hepatitis C.
* ECOG Performance status of 0 or 1.
* Men and women, ≥ 18 years of age. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized.

WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal. Post-menopause is defined as:

* Amenorrhea ≥ 12 consecutive months without another cause, or
* For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level ≥ 35 U/L. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of ipilimumab.

Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study [and for up to 26 weeks after the last doseof investigational product] in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* Evidence of symptomatic CNS lesions as determined by the investigator (patients with asymptomatic lesions or previously irradiated or surgically resected are eligible).
* Any other malignancy from which the patient has been disease-free for less than one year, with the exception of adequately treated basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix.
* Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis).
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
* Patients with ≥ Grade 2 peripheral neuropathy.
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab).
* A history of prior treatment with ipilimumab or prior CD137 agonist or CTLA 4 inhibitor or agonist.
* Concomitant therapy with any of the following: IL 2, interferon, or other non-study immunotherapy regimens; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids.
* Women of childbearing potential (WOCBP), defined above, who:

  1. are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 26 weeks after cessation of study drug, or
  2. have a positive pregnancy test at baseline, or
  3. are pregnant or breastfeeding.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2017-02 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 24 months

SECONDARY OUTCOMES:
Putative Early Cellular and/or Molecular Biomarker levels | 27 months
To determine ORR and clinical benefit rate (ORR + SD ≥ 24 weeks), by immune related response criteria (irRC) and modified WHO criteria (mWHO) of ipilimumab when given with carboplatin and paclitaxel at two different dosing regimens. | 48 months
To determine the overall survival (OS) of patients receiving ipilimumab with carboplatin and paclitaxel. | 48 months
To determine progression free survival (PFS) per irRC and mWHO of patients receiving ipilimumab with carboplatin and paclitaxel. | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Miller, MD, PhD, Principal Investigator — Jewish General Hospital; Rahima Jamal, MD, Principal Investigator — Notre-Dame Hospital (CHUM)
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Jamal R, Lapointe R, Cocolakis E, Thebault P, Kazemi S, Friedmann JE, Dionne J, Cailhier JF, Belanger K, Ayoub JP, Le H, Lambert C, El-Hajjar J, van Kempen LC, Spatz A, Miller WH Jr. Peripheral and local predictive immune signatures identified in a phase II trial of ipilimumab with carboplatin/paclitaxel in unresectable stage III or stage IV melanoma. J Immunother Cancer. 2017 Nov 21;5(1):83. doi: 10.1186/s40425-017-0290-x. PMID 29157311